CLINICAL TRIAL: NCT04841148
Title: A Phase II Trial of Avelumab or Hydroxychloroquine with or Without Palbociclib to Eliminate Dormant Breast Cancer (PALAVY)
Brief Title: Avelumab or Hydroxychloroquine with or Without Palbociclib to Eliminate Dormant Breast Cancer
Acronym: PALAVY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Johns Hopkins University (Other); Translational Breast Cancer Research Consortium (Other); Pfizer (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01121; IRB# 848471 (Other: University of Pennsylvania); TBCRC 046 (Other: Translational Breast Cancer Research Consortium (TBCRC))
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: tumor dormancy; disseminated tumor cells; DTC; minimal residual disease; breast cancer recurrence; CDK4/6 inhibitor; immune checkpoint inhibitor; immunotherapy; autophagy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm, Residual | interventions — Hydroxychloroquine; avelumab; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- HCQ (Experimental): Patients will receive HCQ, 600 mg twice daily D1-28 of each 28-day cycle.
  Interventions: Drug: HCQ
- Avelumab (Experimental): Patients will receive Avelumab, 10 mg/kg, IV, D1 and D15 of each 28-day cycle.
  Interventions: Drug: Avelumab
- Palbociclib and Avelumab (Experimental): Patients will receive Palbociclib 125 mg daily, by mouth on D1-21 concurrently with Avelumab, 10 mg/kg IV on D1 and D15 of each 28-day cycle
  Interventions: Drug: Avelumab; Drug: Palbociclib
- Palbociclib and HCQ (Experimental): Patients will receive Palbociclib 75 mg daily, by mouth on D1-28 concurrently with HCQ, 600 mg twice daily D1-28 of each 28-day cycle.
  Interventions: Drug: HCQ; Drug: Palbociclib

INTERVENTIONS:
Drug: HCQ — 600 mg tablets twice daily D1-28 of each 28-day cycle
  Other Names: Hydroxychloroquine sulfate; Plaquenil
  Arms: HCQ; Palbociclib and HCQ
Drug: Avelumab — 10 mg/kg, IV, D1 and D15 of each 28-day cycle
  Other Names: MSB0010718C; Bavencio
  Arms: Avelumab; Palbociclib and Avelumab
Drug: Palbociclib — 125 mg capsule daily, by mouth on D1-21 concurrently with Avelumab. Or 75 mg capsule daily, by mouth on D1-28 concurrently with HCQ.
  Other Names: Ibrance
  Arms: Palbociclib and Avelumab; Palbociclib and HCQ

SUMMARY:
This clinical trial will assess the safety and early efficacy of Hydroxychloroquine or Avelumab, with or without Palbociclib, in early-stage ER+ breast cancer patients who are found to harbor disseminated tumor cells (DTCs) in the bone marrow after definitive surgery and standard adjuvant therapy.

DETAILED DESCRIPTION:
The overarching goal of this clinical trial is to reduce the incidence of incurable recurrent metastatic breast cancer by targeting the precursors of these recurrences, bone marrow disseminated tumor cells (DTCs) present after definitive treatment. This trial targets unique mechanisms by which DTCs maintain a dormant phenotype (autophagy) and by which they escape dormancy (upregulation of the cyclin-dependent kinase4/6 (CDK4/6) pathway and microenvironmental factors such as immune evasion). The selection of these agents is based upon strong preclinical data demonstrating the relevance of autophagy (inhibited by HCQ), the CDK4/6 pathway (inhibited by palbociclib) and the programmed cell death-1 (PD-1)/Programmed death-ligand 1 (PD-L1) immune checkpoint pathway (blocked by avelumab) as critical mechanisms of cellular and immunological tumor dormancy.

The phase II trial is designed to provide "proof of concept" and estimates of effect of various combinations and durations of these therapies on bone marrow DTCs as a surrogate for ultimate reduction in recurrence. The correlative science aims will provide additional insight into the relationship between the primary tumor and both the biology of DTCs and host immune surveillance for target validation and development, as well as evaluate the role of additional biomarkers both in the bone marrow (with a novel flow-based assay), and in the peripheral circulation (including both circulating tumor cells and cell-free DNA), to identify patients with minimal residual disease (MRD) and targets for intervention and measurement of DTC response.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow aspirate after completion of all definitive therapy demonstrates detectable DTCs (via IHC) as performed by central laboratory assessment at University of Pennsylvania.
* History of stage II-III histologically-confirmed ER+/Her2 neg invasive breast cancer with no evidence of recurrent local or distant disease (by American Joint Committee on Cancer 7th edition). Patients with bilateral breast cancer are eligible, so long as both cancers are ER+/Her2 neg, at least one meets other eligibility criteria and patient is treated with curative intent. For patients who undergo neoadjuvant therapy, eligibility is based upon pathologic stage of residual disease at surgery.
* ER+/Her2 neg receptor status on breast primary tumor (by American Society of Clinical Oncology/College of American Pathologists guidelines). Any partial response (PR) status is allowed. Tumors that are ER negative and PR positive are not eligible. Patients who undergo neoadjuvant therapy are eligible if either the pre-treatment biopsy or residual disease at surgery is ER+/Her2 neg.
* Patients must have completed all primary and adjuvant therapy (including surgery, chemotherapy, and radiation) with the exception of adjuvant endocrine therapy. Prior treatment-related toxicity must be resolved to ≤ Grade 1 with the exception of alopecia and peripheral neuropathy, prior to study enrollment.
* Patients may have received prior CDK4/6 inhibitor therapy with an agent other than Palbociclib. Patients must have discontinued CDK4/6 inhibitor at least 6 months prior to screening.
* Patients must be receiving adjuvant endocrine therapy at the time of enrollment. Patients are eligible to enroll within 2-7 years after initiation of adjuvant endocrine therapy. Use of tamoxifen as adjuvant endocrine therapy during study treatment is not allowed on hydroxychloroquine arms due to the potential drug-drug interaction with hydroxychloroquine. However, patients on tamoxifen at the time of screening may enroll on the treatment trial if switched to an aromatase inhibitor at least 21 days prior to starting study therapy in the event patient is randomized to a hydroxychloroquine containing arm. Premenopausal patients on concurrent ovarian suppression are eligible. Patients on any other adjuvant endocrine therapy, including any investigational therapy, are ineligible.
* Patients receiving bone modifying agents (bisphosphonates or rank-ligand inhibitors) at the time of screening may continue this therapy. Bone modifying agents may not be initiated while receiving study treatment.
* No concurrent enrollment on another investigational therapy clinical trial.
* Men and women, age ≥ 18 years.
* No contraindications to the study medications (refer to Section 7.2) or uncontrolled medical illness.
* Adequate bone marrow, liver, and renal function and other parameters.
* Ability to speak and understand English

Exclusion Criteria:

* Patients with a history of another prior invasive breast cancer are ineligible. Patients with prior Ductal carcinoma in situ (DCIS) of the breast are eligible if this was diagnosed > 5 years prior to enrollment. Patients with prior invasive malignancy other than breast cancer are eligible if they have been disease-free for at least 5 years prior to enrollment.
* Patients receiving chronic, high dose systemic treatment with corticosteroids defined as: chronic use of cortisone >50mg; hydrocortisone >40mg, prednisone >10mg, methylprednisone >8mg or dexamethasone >1.5mg; or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* EKG demonstrating QT interval corrected (QTC) > 480 ms
* Any severe and/or uncontrolled medical conditions or other conditions that could affect subject participation in the study including:

  * Chronic autoimmune disease
  * History or evidence of increased cardiovascular risk including any of the following:

    * Current clinical significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation
    * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrollment
    * Current ≥ Class II congestive heart failure as defined by New York Heart Association
  * History of pneumonitis/interstitial lung disease or severely impaired lung function with a previously documented spirometry and Diffusing Capacity of Lung for Carbon Monoxide (DLCO) that is 50% of the normal predicted value (these tests not required at screening; prior results, if performed for standard of care should be referenced) and/or O2 saturation that is 88% or less at rest on room air
  * Uncontrolled diabetes
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
  * HIV positive patient who are receiving combination anti-retroviral therapy are ineligible because of the potential for pharmacokinetic interactions or increased immunosuppression with Palbociclib. However, HIV per se is not a contraindication to study participation and HIV testing is not required.
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of hydroxychloroquine (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
  * Patients with an active, bleeding diathesis. Patients receiving therapeutic anticoagulation are not eligible for study participation.
  * History of retinopathy or retinal vein occlusion
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of HCQ or Avelumab, alone or in combination with Palbociclib, in eradicating DTCs | Efficacy is assessed at the end of Cycle 6 (each cycle is 28 days).
  Endpoint: Proportion of subjects in each treatment arm with clearance of DTCs at the end of 6 cycles of therapy.

SECONDARY OUTCOMES:
Determine the safety and tolerability of HCQ or Avelumab, alone or in combination with Palbociclib, in this Phase II study: adverse events | Toxicity is assessed from the first dose of study treatment through 30 days after the last dose of study treatment
  Endpoint: Occurrence of an adverse event on treatment by NCI CTCAE v5 criteria.
Estimate the risk of recurrence after treatment with Palbociclib, Avelumab and HCQ, alone or in combination | Recurrence free survival (RFS) will be assessed 3 years after the completion of study treatment
  Endpoint: 3-year recurrence free survival (RFS)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — University of Pennsylvania
Locations (7):
- United States (7):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No